CLINICAL TRIAL: NCT00522223
Title: Sexual Functioning and Quality of Life in Women With Cervical Cancer
Brief Title: Sexual Functioning in Cervical Cancer Survivors
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID02-376; 1R03CA097869-1 (Other: NCI); 1R03CA097869 (NIH)
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Cancer Survivors; Cervix Cancer; Sexual Functioning; Quality Of Life; Questionnaire; Radiation Therapy; Radical Hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire: Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Participants who are treated with radiation therapy: Questionnaires 5 times.
  Participants who undergo a radical hysterectomy: Questionnaires 4 times.
  Other Names: Survey

SUMMARY:
Objectives:

Primary Objectives:

To assess the entire range of sexual functioning (desire, arousal, orgasmic capacity, dyspareunia, and sexual satisfaction) over the course of treatment and early follow-up in patients with local and locally advanced cervical cancer; To assess general cancer-related QOL over the course of treatment and early follow-up in patients with local and locally advanced cervical cancer; To characterize the relationship between sexual dysfunction and overall cancer-related QOL over time; and To identify factors that may predict better sexual function outcomes in patients treated for cervical cancer.

Secondary Objectives:

Describe vaginal changes objectively via measurement of vaginal length. Demonstrate reliability of the vaginal length instrument and its applicability to future studies.

DETAILED DESCRIPTION:
There are two parts to this study. The first part is called a "feasibility study" and will include 20 women who have been treated for cervix cancer in the past. These women will be asked to fill out questionnaires to evaluate their quality of life and sexual functioning. The questionnaires will only be completed once. The questionnaires will be filled out during routine clinic visits.

If the feasibility study is successful (if the majority of the 20 women are able to complete the questionnaires), the second part of the study will be performed with a larger number of women who have been diagnosed with cervix cancer but who have not yet begun treatment. Patients who participate in this part of the study will also be asked to fill out the questionnaires described above.

Participants who are treated with radiation therapy will be asked to complete questionnaires 5 times: before radiation treatment starts, at the time of the first ALTO, and 1 month, 4 months and 7 months after treatment ends. Vaginal measurements will only be done 4 times: at the time of first ALTO, and 1 month, 4 months and 7 months after treatment ends.

Participants who undergo a radical hysterectomy will be asked to complete questionnaires and have a vaginal measurement 4 times: before surgery and 1 month, 4 months and 7 months after treatment ends. Vaginal measurements will only be done 4 times: at the time of first ALTO, and 1 month, 4 months and 7 months after treatment ends.

The questionnaires take about 20 minutes to complete. The vaginal measurement is done by a doctor and takes less than a minute to complete.

This is an investigational study. About 165 patients will take part in this multicenter study. About 135 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility criteria for 20 women in the pilot study (see Treatment Plan for details) of feasibility include: a) History of cervical cancer (within 3 months to 5 years of diagnosis); b) English or Spanish-speaking; and c) Ability to give informed consent.
2. Eligibility criteria for the main study: a) New diagnosis of local or locally advanced cervical cancer; b) English or Spanish-speaking; and c) Ability to give informed consent.

Exclusion Criteria:

1. Patients who are illiterate.
2. Patients who have undergone an exenteration.
3. Patients who do not speak English or Spanish.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with history of cervical cancer.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2002-09-10 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
To evaluate sexual functioning and the quality of life (QOL) in women with cervix cancer. | 7 Years

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org